CLINICAL TRIAL: NCT03716115
Title: Therapeutic Approaches to Malnutrition Enteropathy: Phase II Trials of Four Novel Interventions in Children in Zambia and Zimbabwe
Brief Title: Therapeutic Approaches to Malnutrition Enteropathy
Acronym: TAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 011724 QM
Record Dates: First submitted 2018-10-08; First posted 2018-10-23 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2018-09

CONDITIONS: Severe Acute Malnutrition
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Acetylglucosamine; teduglutide; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Colostrum (Experimental): Colostrum high protein powder (Neovite) given orally or through NG tube 1.5g daily, in addition to standard care following WHO guidelines for management of SAM.
  Interventions: Dietary Supplement: Colostrum high protein powder (Neovite)
- GInNAC (Experimental): N-Acetyl glucosamine (GInNAC). Given orally (1g three times daily) for 14 days, gradually increased from 0.5g to avoid osmotic diarrhoea, in addition to standard care following WHO guidelines for management of SAM.
  Interventions: Drug: N-Acetyl Glucosamine (GInNAC)
- Teduglutide (Experimental): Teduglutide s/c. Administration by subcutaneous injection (0.5mg/kg/day) daily for 14 days, in addition to standard care following WHO guidelines for management of SAM.
  Interventions: Drug: Teduglutide
- Budenoside (Experimental): Budesonide 3mg orally daily for 14 days, then rapidly tapered, in addition to standard care following WHO guidelines for management of SAM.
  Interventions: Drug: Budesonide
- Standard care (No Intervention): Standard care following WHO guidelines for management of SAM.

INTERVENTIONS:
Dietary Supplement: Colostrum high protein powder (Neovite) — Bovine colostrum provided as powder will be reconstituted and administered orally or via NG tube.
  Arms: Colostrum
Drug: N-Acetyl Glucosamine (GInNAC) — N-Acetyl glucosamine provided as powder will be reconstituted and administered orally or via NG tube.
  Arms: GInNAC
Drug: Teduglutide — Teduglutide will be administered daily as subcutaneous injection
  Arms: Teduglutide
Drug: Budesonide — Budesonide liquid (as marketed for nebulisation) will be administered orally or bia NG tube daily.
  Arms: Budenoside

SUMMARY:
The TAME study will evaluate four new approaches which will be compared against the standard care currently in use in the treatment of malnutrition enteropathy in children with severe acute malnutrition. A high pathogen burden causes damage to the intestinal mucosa which exacerbates nutritional impairment and leads to further susceptibility to infection and impaired epithelial regeneration. Enteropathy is characterised by multiple epithelial breaches, microbial translocation from gut lumen to systemic circulation and systemic inflammation.The trial will evaluate the potential impact of four interventions (colostrum, N-acetyl glucosamine, teduglutide, and budesonide) given for 14 days, which aim at mucosal restoration. The trial will determine if repairing damage to the small intestinal mucosa leads to the reduction of systemic inflammation and thus lessening the nutritional impairment, and so if this contributes to the reduction of mortality in children.

In Zambia only, endoscopic biopsies and confocal laser endomicroscopy will be used to evaluate response and confirm safety at a mucosal level.

Identifying an agent or agents which contribute most to mucosal healing will then ultimately lead to further large phase 3 trial in which the agent(s) will be further evaluated.

The trial also anticipates to gain a more in depth understanding of pathophysiology and may identify where current management strategies of treating malnutrition enteropathy in children are failing.

DETAILED DESCRIPTION:
Over the last two decades, three key developments in the approach to treatment have improved the outcome of SAM: standardised management protocols, ready to use therapeutic food (RUTF), and community management of acute malnutrition (CMAM). CMAM has four components, namely, community mobilization and community identification of cases of acute malnutrition, supplementary feeding programme (SFP) for children with moderate acute malnutrition (MAM), outpatient therapeutic programme (OTP) of SAM with no medical complications and inpatient management of SAM with medical complications However, severely malnourished children with medical complications requiring hospitalisation often fail to respond to treatment, and continue to experience high inpatient mortality of up to 35%. Even after discharge, children have a poor prognosis, with 42% mortality over the subsequent year. It is a subgroup of children with SAM and acute or persistent diarrhoea who pose the most difficult management challenges, although the vast majority of children with SAM have substantial degree of enteropathy. Current treatment guidelines for SAM are not well supported by an evidence base, and there is a dearth of clinical trial data; in particular, there are no specific interventions to target enteropathy in SAM. In a systematic review, only three trials were found which inform management of SAM and persistent diarrhoea, and no trials dealing with the HIV-infected child. The investigators therefore believe that novel therapeutic approaches are urgently needed, and that a series of small phase 2 trials could guide development of a new generation of treatments. These trials should focus on repairing damage to the small intestinal mucosa, as there is now substantial evidence that this plays a central role in the genesis of systemic inflammation, bacterial translocation and sepsis with all its adverse nutritional consequences.

Evidence of malnutrition enteropathy: Recent studies have been highly informative about the infectious contribution to dysfunction of the small intestine in malnourished children. A high pathogen burden causes damage to the mucosa which exacerbates nutritional impairment and leads to further susceptibility to infection and impaired epithelial regeneration, in a cyclical process first described in Central America in the 1970s. This mucosal damage in SAM is here referred to as malnutrition enteropathy. In previous studies, markers of microbial translocation and systemic inflammation were dramatically increased in children with SAM compared to healthy controls. Enteropathy is characterised by multiple epithelial breaches, microbial translocation from the gut lumen to the systemic circulation, and systemic inflammation. Epithelial breaches were present in histological (haematoxylin/eosin-stained) sections and sections studies using immunofluorescence for claudin 4 and E-cadherin. In adults, these lesions were shown to occur in vivo using confocal laser endomicroscopy. There was also a consistent pattern of blunted epithelial repair, with reduced glucagon-like peptide 2 (GLP2) in serum, reduced trefoil factor 3 in duodenal aspirates, and a strong transcriptomic signature of impaired mucosal defence. Two further immunological abnormalities were identified in children with malnutrition enteropathy: low-level false positive coeliac-like autoantibodies, and upregulation of SMAD7 similar to the pattern seen in Crohn's disease. Together, these abnormalities indicate there is substantial structural and functional damage to the small intestine, and that this primary gut pathology is associated with systemic sequelae.

WHO guidelines clearly state that antibiotic treatment should be part of the initial management of all cases of SAM, whether associated with overt features of infection ('complicated' SAM) or not ('uncomplicated' SAM). Antibiotic use was associated with reduced short term mortality and improved nutritional rehabilitation in SAM with no medical complications in Malawi but post-discharge prophylaxis with cotrimoxazole did not reduce long-term mortality following complicated SAM in Kenya, and in Niger antibiotics conferred no benefit. Even in the best outcome group in the Malawi antibiotic trial, mortality was not reduced below 4% over 12 weeks in children managed as outpatients in OTP. This seems to be a glass floor below which it has never been possible to reduce mortality in SAM, even in uncomplicated cases in the community or in clinical trials. In SAM with medical complications who are managed as inpatients, mortality is much higher, and when combined with HIV infection can reach 35% in hospital and 62% over one year post-discharge.

If optimal antibiotics are insufficient to reduce mortality below 4% in uncomplicated cases treated in the community, and mortality is much higher in complicated cases, there must be other factors which lead inexorably to adverse outcomes in a subgroup of children with complicated SAM. It seems that a major contributor to the residual mortality observed after current optimal therapies have been implemented is failure of restitution in the gut. This means that in a subset of children with SAM, largely but not exclusively those with persistent diarrhoea, the intestinal mucosa is damaged and leaky, permitting efflux of plasma proteins and influx of luminal microbial products, and fails to repair following the infective insult. The evidence leading to this interpretation is:

i. In children with SAM and persistent diarrhoea, there are epithelial gaps visualised in haematoxylin/eosin-stained sections and using immunohistochemistry for claudin-4 and E-cadherin; ii. These are morphologically similar to lesions seen in environmental enteropathy in adults, though more severe and more numerous; iii. Plasma proteins are easily detected in western blots of duodenal aspirates, suggesting leakage from blood to gut lumen; iv. Biomarkers of microbial products (bacterial DNA and lipopolysaccharide) are found in very high concentrations in peripheral blood, direct evidence of microbial translocation from lumen to blood; v. Children with persistent diarrhoea and malnutrition have reduced circulating concentrations of glucagon-like peptide-2 (GLP2) and reduced trefoil factor 3 in intestinal secretions, suggesting a failure of homeostatic repair mechanisms. Circulating LPS was inversely proportional to circulating GLP2, and this remained true in multivariate analysis.

In a recent study of children with complicated SAM in Malawi, children who died were more likely to have diarrhoea and higher levels of faecal calprotectin (a marker of intestinal inflammation), and levels of systemic inflammation were directly related to mortality. There is now clear evidence that enteropathy is associated with systemic inflammation and mortality in SAM and a new treatment paradigm is required to improve outcomes.

There is a need for new approaches. The investigators postulate that the central lesion in malnutrition enteropathy is epithelial leakiness through tight junction damage and microerosions, and so propose therapy directed at restoration of the mucosal barrier which will permit reversal of the cascade of downstream inflammatory derangements. Novel approaches are required in order to achieve a radical improvement in outcome, and reduce current unacceptably high mortality rates. The TAME trial will investigate four potential therapeutic approaches to achieving mucosal restoration. Colostrum, teduglutide and N-acetyl glucosamine are all intended to achieve mucosal healing. Budesonide, a corticosteroid with limited absorption, is targeted at the downstream inflammatory changes; in inflammatory conditions such as coeliac disease or Crohn's disease, steroids produce rapid clinical response. If any of these interventions impact on malnutrition enteropathy, it will become possible to trial these novel therapeutic approaches in phase 3 trials to detect an impact on our world's most disadvantaged children. The trial will also generate useful information about pathophysiology.

The novel therapeutic approaches to be tested in the TAME trial are:

* Colostrum: high-protein bovine colostrum powder (Neovite) orally 1.5 g every 8 hours for 14 days, reconstituted with water and given through a nasogastric (NG) tube or orally. Colostrum reduces the increased epithelial permeability seen in heat shock. Colostrum contains nutrients, immunoglobulins and growth factors, including epidermal growth factor (EGF) and insulin-like growth factor 1 (IGF-1).
* N-acetyl glucosamine (GlcNAc) will be given orally or via NG tube for 14 days, gradually increased from a starting dose of 0.5g, to 1g three times daily to avoid osmotic diarrhoea. Impaired glycosylation of glycosaminoglycans has been noted in oedematous malnutrition, with reduced concentrations of glycosaminoglycans found in blood, urine, kidney, brain and small intestine. Specific consequences of reduced heparan sulphate expression include gut epithelial leakiness with hypoalbuminaemia. GlcNAc administration has been demonstrated to restore the intestinal epithelial charged barrier in Crohn's disease. GlcNAc may theoretically induce osmotic diarrhoea if not absorbed in the small intestine. Although this has not been observed clinically in animals or in older children we will use a dose escalation schedule to minimise the chance of this.
* Teduglutide by subcutaneous injection (0.05mg/kg/day) daily for 14 days. Teduglutide is a long-acting form of GLP2 which has proven efficacy in intestinal failure, improving absorption and reducing the need for parenteral support. GLP2 is a hormone secreted by L cells in the terminal ileum, which drives epithelial repair and mediates intestinal adaptation by increased cellular proliferation and villus hypertrophy.
* Budesonide 3mg orally daily for 7 days, then 2mg for 4 days then 1mg for 3 days. Budesonide is standard therapy for Crohn's disease, and can be used for refractory coeliac disease. Since malnutrition enteropathy is characterized by intestinal inflammation, with infiltration of activated T cells, an anti-inflammatory approach is rational. A prior trial of mesalazine in Kenya confirmed an immuno-modulatory approach is safe in the setting of SAM, but targeting the small, rather than large, intestine with a more potent agent is likely to be more effective.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6 - 59 months, of either sex;
2. Inpatient in the paediatric wards of one of the research sites;
3. Hospitalised with Severe Acute Malnutrition (SAM, defined using WHO definition: weight-for-length z score of less than -3, or mid upper arm circumference of less than 11.5cm, and/or bilateral pedal oedema);
4. Clinically stable*;
5. With written, informed consent from the primary caregiver(s); the child cannot be enrolled if the primary caregiver(s) cannot give consent.

   * Judged by the medical team on a case by case basis, but in general a child without shock, hypothermia, hypoglycaemia or reduced conscious level.

Exclusion Criteria:

1. Clinically unstable*;
2. Less than 5kg body weight;
3. Neurological disability which would explain or partly explain poor feeding;
4. Oro-facial abnormalities which would explain or partly explain poor feeding;
5. Caregiver unwilling to consent to child HIV testing;
6. Haemoglobin concentration < 6 g/dl at the time of enrolment;
7. Caregiver unwilling to remain in hospital for the duration of the study treatment;
8. Any underlying condition, other than HIV, which in the opinion of the investigator would put the subject at undue risk of failing study completion or would interfere with analysis of study results;
9. Contraindication to any of the trial treatments (e.g. allergy to cow's milk protein).

   * As assessed by the medical team on a case-by-case basis, but in general a clinically unstable state would include shock, hypothermia, hypoglycaemia or reduced conscious level.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Composite measure of concentration of three faecal inflammatory markers | 14-18 days
  Composite measure of concentration of three faecal inflammatory markers (myeloperoxidase, neopterin, alpha1-antitrypsin) measured by ELISA

SECONDARY OUTCOMES:
Lactulose:rhamnose ratio | 14-18 days
  Lactulose:rhamnose ratio of concentration in urine samples collected over 2 hours following oral administration of test dose
Plasma lipopolysaccharide (LPS) | 14-18 days
  Plasma LPS concentration measured by limulus amoebacyte lysate assay
Plasma biomarker lipopolysaccharide binding protein (LBP) | 14-18 days
  Plasma LBP concentration measured by ELISA
Plasma fatty acid binding protein (FABP) | 14-18 days
  Plasma FABP concentration measured by ELISA
Plasma soluble CD14 | 14-18 days
  Plasma concentration of soluble CD14 measured by ELISA
Plasma CD163 | 14-18 days
  Plasma concentration of CD163 measured by ELISA
Plasma CRP | 14-18 days
  Plasma concentration of C-reactive protein measured by ELISA
Plasma albumin | 14-18 days
  Plasma concentration of albumin measured by ELISA
Mortality | 14 days and 28 days
  Number of deaths in each treatment allocation group
Adverse events | 14 days and 28 days
  Number of adverse events in each treatment allocation group
Change in weight and length | 14 days and 28 days
  Change in weight and length measured by experienced nurses and expressed as change in weight-for-length z score compared to WHO standard
Days with diarrhoea | 14-18 days
  Number of days during which diarrhoea was experienced assessed by experienced nurses
Days with fever | 14-18 days
  xv. Days with fever (two or more recordings of core temperature of 37.8oC or higher in any 24 h period)
Villus height: crypt depth ratio | 14-18 days
  Change in villus height and crypt depth measured in endoscopic biopsies (Lusaka only)
Epithelial leakiness | 14-18 days
  Leakage of fluorescein into gut lumen assessed by Watson score during confocal laser endomicroscopy (Lusaka only)
Tertiary Objectives-Tertiary Endpoints- Exploratory work on glyscosylation | 14-18 days
  Glycosylation in saliva and biopsies

OTHER OUTCOMES:
Metabolomics | 14-18 days
  Untargeted metabolomic profile by mass spectroscopy, and specific measurement of citrulline, tryptophan and kynurenine
Transcriptomic analysis | 14-18 days
  Untargeted analysis of mRNA sequencing data from intestinal biopsies
Confocal laser endomicroscopy | 14-18 days
  Mucosal leakiness measured by observation of plumes and luminal fluorescein during confocal laser endomicroscopy
Biomarker concentrations | 14-18 days
  Inflammatory markers: CCL3, CCL4, CCL11, GCSF, GM-CSF, IFN-gamma, IL-1b, IL-1ra,IL2, IL-6, IL-8, IL-10, IL-33, TNF-a Endothelial markers: Angiopoetin-1, D-dimer, EGF, ICAM1, IGFBP-3, PIGF, CD62L, CD62P, TPO, VCAM1, VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kelly, MD, Study Chair — Queen Mary University of London; Beatrice Amadi, MD, Principal Investigator — University Teaching Hospital, Lusaka, Zambia; Andrew Prendergast, PhD, Principal Investigator — Queen Mary University of London; Mutsa Bwakura-Dangarembizi, MB, Principal Investigator — Parirenyatwa Hospital, Harare, Zimbabwe
Locations (3):
- University Teaching Hospital, Nationalist Road, Lusaka, Zambia
- Zimbabwe (2):
  - Harare Central Hospital, Harare
  - Parirenyatwa Hospital, Harare

REFERENCES:
- [Derived] Chandwe K, Bwakura-Dangarembizi M, Amadi B, Tawodzera G, Ngosa D, Dzikiti A, Chulu N, Makuyana R, Zyambo K, Mutasa K, Mulenga C, Besa E, Sturgeon JP, Mudzingwa S, Simunyola B, Kazhila L, Zyambo M, Sonkwe H, Mutasa B, Chipunza M, Sauramba V, Langhaug L, Mudenda V, Murch SH, Hill S, Playford RJ, VanBuskirk K, Prendergast AJ, Kelly P. Malnutrition enteropathy in Zambian and Zimbabwean children with severe acute malnutrition: A multi-arm randomized phase II trial. Nat Commun. 2024 Apr 17;15(1):2910. doi: 10.1038/s41467-024-45528-0. PMID 38632262
- [Derived] Kelly P, Bell L, Amadi B, Bwakura-Dangarembizi M, VanBuskirk K, Chandwe K, Chipunza M, Ngosa D, Chulu N, Hill S, Murch S, Playford R, Prendergast A. TAME trial: a multi-arm phase II randomised trial of four novel interventions for malnutrition enteropathy in Zambia and Zimbabwe - a study protocol. BMJ Open. 2019 Nov 14;9(11):e027548. doi: 10.1136/bmjopen-2018-027548. PMID 31727642